CLINICAL TRIAL: NCT07076407
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled, Multicenter Study to Evaluate Azetukalner in Moderate-to-Severe Major Depressive Disorder
Brief Title: A Randomized Study of Azetukalner Versus Placebo in Major Depressive Disorder (X-NOVA3)
Acronym: X-NOVA3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPF-010-D302
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Antidepressant; XEN1101; Azetukalner
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azetukalner (Experimental): Azetukalner 20 mg
  Interventions: Drug: Azetukalner
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azetukalner — Azetukalner 20 mg taken orally once a day with food (with the evening meal when possible) for 6 weeks
  Other Names: XEN1101
  Arms: Azetukalner
Drug: Placebo — Placebo taken orally once a day with food (with the evening meal when possible) for 6 weeks
  Arms: Placebo

SUMMARY:
X-NOVA3 is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the clinical efficacy, safety, and tolerability of azetukalner as a monotherapy in adult participants diagnosed with Major Depressive Disorder (MDD)

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥18 and ≤74 years of age and experienced their first major depressive episode (MDE) prior to 50 years of age
* Body Mass Index (BMI) ≤40 kg/m2
* Meets the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition Text Revised (DSM-5-TR) criteria for current major depressive disorder and is currently in an MDE, confirmed using the Mini International Neuropsychiatric Interview (MINI)
* Participant's current MDE has a duration of ≥6 weeks and ≤24 months.

Key Exclusion Criteria:

* Participant has a primary diagnosis of a mood disorder other than MDD.
* Participant has a history of any of the following: MDD with psychotic or catatonic features; MDD with mixed features; Bipolar I or II disorder; Obsessive-compulsive disorder; Schizophrenia, primary thought disorder, or other psychotic disorder.
* Participant has a current diagnosis of any of the following: MDD with seasonal pattern; Depression with peripartum or perimenopausal onset; Post traumatic stress disorder; Antisocial or borderline personality disorder (or presence of clinically significant borderline personality traits); Panic disorder and/or agoraphobia; ADHD treated with a psychostimulant, diagnosed during the current MDE, or with unstable symptoms, as judged by the investigator.
* Participant has a substance (excluding tobacco) or alcohol use disorder within the 12 months prior to screening.
* Participant has had an active suicidal plan/intent within the 6 months prior to screening, presence of suicidal behavior in the last 2 years, or >1 suicide attempt > 24 years of age.
* Participant has a history of non-suicidal self-harm behavior in the 12 months prior to screening.
* Participant has used antidepressants or other prohibited medications (including benzodiazepines), within the 2 weeks (4 weeks for fluoxetine) or within a period less than 5 times the drug's half-life, whichever is longer, prior to randomization.
* Participant has a history of non-response to ≥2 antidepressant drugs of adequate dose and duration in the current MDE as determined by the Antidepressant Treatment Response Questionnaire (ATRQ).
* Participants with medical conditions that may interfere with the purpose or conduct of the study
* Participant is pregnant, breastfeeding, or planning to become pregnant.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Hamilton Depression Rating Scale, 17-item (HAMD-17) score at Week 6 | Baseline to Week 6
  The HAMD-17 consists of 17 items that are used to rate the severity of depression symptoms. Each item is scored in a range of 0 to 2 points or 0 to 4 points, with higher scores indicating a greater degree of depression. The score for each item is summed to compute a total score, which ranges from 0 to 52 points.

SECONDARY OUTCOMES:
Change from baseline in the Snaith-Hamilton Pleasure Scale (SHAPS) score at Week 6 | Baseline to Week 6
  The SHAPS is a 14-item self-report questionnaire used to assess anhedonia. Each item on the SHAPS is worded so that higher scores indicate greater anhedonia. A total score can be derived by summing the responses to each item. Items answered with "strongly agree" are assigned a score of 1, while "strongly disagree" responses are assigned a score of 4 points. Total scores on the SHAPS can range from 14 to 56 points, with higher scores corresponding to higher levels of anhedonia.
Change from baseline in the Hamilton Depression Rating Scale, 17-item (HAMD-17) score at Week 1 | Baseline to Week 1
  The HAMD-17 consists of 17 items that are used to rate the severity of depression symptoms. Each item is scored in a range of 0 to 2 points or 0 to 4 points, with higher scores indicating a greater degree of depression. The score for each item is summed to compute a total score, which ranges from 0 to 52 points.
Change from baseline in the Clinical Global Impression of Severity (CGI-S) score at Week 6 | Baseline to Week 6
  The CGI-S is a clinician-rated global measure of participant overall disease severity. Participants are rated on a 7-point severity scale, with higher scores indicating more severe depression.
To assess the safety and tolerability of azetukalner (e.g., adverse events) | From screening (approximately 4 weeks prior to baseline) through to 8 weeks post-final dose.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - University of Alabama at Birmingham, Huntsville Regional Medical Campus, Huntsville, Alabama
  - Pillar Clinical Research, Bentonville, Arkansas
  - SanRo Clinical Research Group, Bryant, Arkansas
  - Clinical Innovations Inc, Bellflower, California
  - Center for Neurohealth, La Jolla, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Neuroscience Research, Sherman Oaks, California
  - Pacific Clinical Research Management Group, Upland, California
  - Institute of Living, Hartford, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Equipath Health and Research Tampa Bay, Llc, Riverview, Florida
  - Delricht Research, Atlanta, Georgia
  - Advanced Quality Medical Research, Orland Park, Illinois
  - Pharmasite Research Inc., Baltimore, Maryland
  - Adams Clinical Boston, Boston, Massachusetts
  - Activmed Practices & Research, Llc - Methuen, Methuen, Massachusetts
  - Adams Clinical Watertown, Watertown, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Fieve Clinical Research, Inc., New York, New York
  - Magnolia Clinical Research, Llc, Cary, North Carolina
  - Insight Clinical Trials, Independence, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Austin Clinical Trial Partners, Austin, Texas
  - Boeson Research, Provo, Utah

IPD SHARING:
Plan to Share IPD: No